CLINICAL TRIAL: NCT04974658
Title: Analgesic Efficacy of the Novel Intra- Semispinal Fascial Plane Block in Posterior Cervical Spine Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Naglaa Fathy Abdelhaleem Abdelhaleem, Lecturer, Anesthesia and Surgical Intensive Care department, Faculty of Medicine, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: #6955
Record Dates: First submitted 2021-07-14; First posted 2021-07-23 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Cervical Spine Surgery
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: This study will be performed in neurosurgical operating rooms at Zagazig University Hospitals and included 52 patients allocated randomly into two groups: 26 patients recruited in the block group (I) for the Inter-semispinal plane block and 26 patients recruited in the (C) control group.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Randomization assignments will be kept in sealed envelopes until all preprocedural measurements will be completed, and then they are opened by the research anesthesiologist immediately prior to the nerve block.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The block group (ISP) (Active Comparator): After aseptic preparation of the injection area, the needle will be introduced in-plane through the skin and advanced into the fascial plane between the semispinalis cervicis and semispinalis capitis muscles. After negative aspiration for blood, 20 ml of 0.25% bupivacaine on each side will be injected for each block.
  Interventions: Procedure: Inter-semispinal plane block
- control group (C) (Placebo Comparator): No block will be performed
  Interventions: Procedure: Inter-semispinal plane block

INTERVENTIONS:
Procedure: Inter-semispinal plane block — Ultrasound Inter-semispinal plane block in block group
  Other Names: No block intervention in control group

SUMMARY:
Posterior cervical spine surgery often requires a large posterior midline incision, resulting in poorly controlled postoperative pain, which arises from iatrogenic mechanical damage, intraoperative retraction, and resection to structures such as bone, ligaments, muscles, intervertebral discs, and zygapophysial joints.

DETAILED DESCRIPTION:
Ultrasound-guided Inter-semispinal plane (ISP) block, was proposed as a novel technique for analgesia in posterior cervical spine surgeries. The ISP block involves an injection of local anesthetic into the fascial plane between the semispinalis cervicis and semispinal capitis muscles and results in blocking the dorsal rami of the cervical spinal nerves. ISP block can provide effective analgesia in posterior cervical spine surgery

ELIGIBILITY:
Inclusion Criteria:

* Patients' acceptance.
* ASA I , II andIII .
* Age between 18 years up to 70 years in both sexes.
* Patients with a BMI (body mass index) ranging from 18.5 to 30 kg/m2.
* Patients who scheduled for elective posterior cervical spine surgeries

Exclusion Criteria:

* Uncooperative patients
* Coagulopathy.
* Local tissue infection.
* Allergy to local anesthesia.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2021-08-10 (Actual); Primary Completion 2022-07-11 (Actual); Study Completion 2022-07-11 (Actual)

PRIMARY OUTCOMES:
Total morphine consumed for 24 hours postoperative will be calculated. | Total morphine consumed up to 24 hours postoperative
  Calculation of total morphine that will be used postoperatively. Postoperative morphine will be considered if the postoperative VAS score >3 or the patient requested additional analgesia. Rescue analgesia of intravenous morphine will be given

SECONDARY OUTCOMES:
Total fentanyl consumed intraoperative will be calculated | total fentanyl dose that will be used for entire operative time.
  Total intraoperative fentanyl consumption including the induction doses (1mic/ kg) plus the additional doses of fentanyl (from 0.5 to 1 mic) that will be given if heart rate or blood pressure increases above 20%.
postoperative pain will be assessed using the Numerical Pain Score (NRS) score | NRS will be recorded 24 hours postoperative.
  Numerical Pain Score (NRS) ranges from 0 to 10, where 0 is no pain, and 10 is the worst pain imaginable. Adequate pain control will be considered at Numerical Pain Score (NRS) < 4.

CONTACTS AND LOCATIONS:
Overall Officials: Naglaa F Abdelhaleem, MD, Principal Investigator — Faculty of medicine, Zagazig University Hospitals
Locations (2):
- Egypt (2):
  - Faculty of Medicine, Zagazig University, Zagazig
  - Faculty of medicine, Zagazig

IPD SHARING:
Plan to Share IPD: Yes
Data will be available on permission
Supporting Information: Study Protocol, SAP
Time Frame: After one year from publishing to a journal

REFERENCES:
- [Background] Ohgoshi Y, Kubo EN. Inter-semispinal plane block for cervical spine surgery. J Clin Anesth. 2018 May;46:94-95. doi: 10.1016/j.jclinane.2018.02.007. Epub 2018 Feb 9. No abstract available. PMID 29433034